CLINICAL TRIAL: NCT00553969
Title: Efficacy of Coreg CR and Lisinopril on Markers for Cardiovascular Functional and Structural Disease. DETECT (DEtection and Treatment of Early Cardiovascular Disease Trial)
Brief Title: Efficacy of Coreg CR and Lisinopril on Markers for Cardiovascular Functional and Structural Disease
Acronym: DETECT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0709M15829
Record Dates: First submitted 2007-11-05; First posted 2007-11-06 (Estimated); Results first posted 2014-12-17 (Estimated); Last update posted 2018-04-24 (Actual); Status verified 2018-03

CONDITIONS: Pre-hypertension
Keywords: cardiovascular disease prevention
MeSH Terms: conditions — Prehypertension | interventions — Carvedilol; Lisinopril

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): Coreg CR + lisinopril
  Interventions: Drug: carvedilol phosphate and lisinopril
- 2 (Experimental): Coreg CR + placebo
  Interventions: Drug: carvedilol phosphate
- 3 (Experimental): lisinopril + placebo
  Interventions: Drug: lisinopril
- 4 (Placebo Comparator): placebo + placebo
  Interventions: Drug: placebo and placebo

INTERVENTIONS:
Drug: carvedilol phosphate — Extended release capsules, 20mg once daily for 1 month, 40mg once daily for 8 months
  Other Names: Coreg CR
  Arms: 2
Drug: lisinopril — tablets, 10mg once daily for 1 month, 20mg once daily for 8 months
  Arms: 3
Drug: carvedilol phosphate and lisinopril — carvedilol phosphate = extended release capsules, 20mg once daily for 1 month, 40mg once daily for 8 months; lisinopril= tablets, 10mg once daily for 1 month, 20mg once daily for 8 months
  Other Names: Coreg CR (carvedilol phosphate)
  Arms: 1
Drug: placebo and placebo — capsule once daily for 9 months; dosage unknown
  Arms: 4

SUMMARY:
This study will examine the individual and combined effects of Coreg CR and lisinopril, on cardiovascular health as measured by Rasmussen Disease Score (RDS) in a blinded, placebo controlled comparison over a 9-month study period. Patients to be randomized will have pre-hypertensive blood pressures that do not require anti-hypertensive therapy and at least one additional cardiovascular risk factor.

DETAILED DESCRIPTION:
* This study will compare the effect of Coreg CR and lisinopril, separately and together, on Rasmussen Disease Score in a controlled study with an inactive substance (placebo).
* Study patients will have pre-hypertensive (slightly elevated) blood pressures not requiring therapy.
* Lisinopril is an angiotensin converting enzyme (ACE) inhibitor. Angiotensin is a chemical that is made by the body continuously. Angiotensin narrows blood vessels and thereby maintains (elevates) blood pressure. When the enzyme is blocked by lisinopril, angiotensin cannot be converted into its active form. As a result, blood pressure is lowered. Lisinopril is a drug that has been approved for use by the U.S. Food and Drug Administration (FDA) and health authorities for the treatment of high blood pressure and heart failure.
* Coreg CR is a once-a-day heart medication that is part of a class of drugs known as beta-blockers. Beta-blockers prevent beta-adrenergic substances such as adrenaline from activating parts of the nervous system, including the heart. Beta-blockers therefore relieve stress on the heart by slowing heart beat, decreasing the force of heart muscle contractions, and reducing blood pressure. Coreg has also been approved by the FDA for the treatment of hypertension and various other cardiovascular conditions.
* It is possible that the beta blocker could increase the benefits of the ACE inhibitor by inhibiting renin production, which is an important step in angiotensin production. These two drugs may act together to provide even more protection to blood vessels and the heart.

ELIGIBILITY:
Inclusion Criteria:

* Males and females > 18 years old with pre-hypertensive or borderline blood pressures (systolic blood pressure ≥ 130 mmHg or diastolic blood pressure ≥ 85 mmHg) deemed not to need antihypertensive therapy. Subjects must also have one additional risk factor for cardiovascular disease, including:
* LDL > 130 and < 160 mg/dL
* HDL < 40 mg/dL
* Fasting blood sugar >100 and < 126 mg/dL
* Body mass index ≥ 30
* Smoker
* Family history of premature heart disease or hypertension

Exclusion Criteria:

* Patients with a history of cardiac, cerebral or other vascular events within the previous 6 months will be excluded. Other exclusions include background therapy with a beta blocker or ACE inhibitor therapy, known or suspected intolerance to beta blockers or ACE inhibitors, angiotensin receptor blocker therapy, or diabetes. Pregnant or lactating women, and women of child-bearing age who are not using an acceptable form of contraception are also excluded from this study.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2007-11; Primary Completion 2010-09 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jay N Cohn, MD, Principal Investigator — Professor, University of Minnesota, Cardiology Division
Locations (1):
- University of Minnesota, Variety Club Research Center 102, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- 1 Coreg CR + Lisinopril: Coreg CR + lisinopril
  carvedilol phosphate and lisinopril : carvedilol phosphate = extended release capsules, 20mg once daily for 1 month, 40mg once daily for 8 months; lisinopril= tablets, 10mg once daily for 1 month, 20mg once daily for 8 months
- 2 Coreg CR + Placebo: Coreg CR + placebo
  carvedilol phosphate : Extended release capsules, 20mg once daily for 1 month, 40mg once daily for 8 months
- 3 Lisinopril + Placebo: lisinopril + placebo
  lisinopril : tablets, 10mg once daily for 1 month, 20mg once daily for 8 months
Period: Overall Study
Arm/Group | 1 Coreg CR + Lisinopril | 2 Coreg CR + Placebo | 3 Lisinopril + Placebo | 4 Placebo + Placebo
Started | 31 | 24 | 22 | 24
Completed | 23 | 24 | 21 | 23
Not Completed | 8 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 Coreg CR + Lisinopril | 2 Coreg CR + Placebo | 3 Lisinopril + Placebo | 4 Placebo + Placebo | Total
Number analyzed (Participants) | 23 | 24 | 21 | 23 | 91
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 23 | 24 | 21 | 23 | 91
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (13) | 53 (10) | 53 (10) | 51 (13) | 52.25 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 5 | 8 | 26
  Male | 17 | 17 | 16 | 15 | 65
Region of Enrollment [Number; unit: participants]
  United States | 23 | 24 | 21 | 23 | 91

OUTCOME MEASURES:

1. Primary Outcome: Change in Disease Score (DS) Among the Treatment Groups
Description: Rasmussen Disease Score (RDS) Change From Baseline to 9 Months A score of six or higher on these tests means the patient likely has plaque build-up in the arteries, or atherosclerosis, while a score of three to five suggests that such a problem may be developing. A score of two or less signals a patient is fine but should return in the future for another test. The method detects disease at the earliest moment, before the traditionally used calcium score would show any signs of trouble.
Time Frame: Baseline and nine months
Population: Calculation for change is the value at the later time point minus the value at the earlier time point.
Measure: Mean (Standard Deviation); unit: Overall Rasmussen Disease Score Change
Arm/Group | 1 Coreg CR + Lisinopril | 2 Coreg CR + Placebo | 3 Lisinopril + Placebo | 4 Placebo + Placebo
Number analyzed (Participants) | 23 | 24 | 21 | 23
Overall Rasmussen Disease Score Change | -2.48 (1.9) | -2.29 (2.3) | -2.38 (2.6) | -0.96 (1.5)

ADVERSE EVENTS:
Arm/Group | 1 Coreg CR + Lisinopril | 2 Coreg CR + Placebo | 3 Lisinopril + Placebo | 4 Placebo + Placebo
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/24 | 1/22 | 0/24
Other Adverse Events (participants affected / at risk) | 0/31 | 0/24 | 0/22 | 0/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 1 Coreg CR + Lisinopril (N=31) | 2 Coreg CR + Placebo (N=24) | 3 Lisinopril + Placebo (N=22) | 4 Placebo + Placebo (N=24)
stroke (Vascular disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No